CLINICAL TRIAL: NCT04712786
Title: Refractive Changes in Pseudophakic Eyes Following Vitrectomy With or Without Gas Tamponade
Brief Title: Refractive Changes Following Vitrectomy
Status: Completed | Type: Observational
Sponsor: Bursa Retina Eye Hospital (Other)
Responsible Party: Principal Investigator, sami yilmaz, Medical doctor, ophthalmology specialist, Bursa Retina Eye Hospital
Other Study IDs: BursaRetinaEyeH
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Retinal Detachment; Refractive Errors; Vitreous Hemorrhage; Epiretinal Membrane
Keywords: Myopic shift; Gas tamponade; Pars plana vitrectomy
MeSH Terms: conditions — Retinal Detachment; Refractive Errors; Vitreous Hemorrhage; Epiretinal Membrane

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group: 27 patients, Group 1 consisted of patients with pseudophakic rhegmatogoneous retinal detachment who underwent pars plana vitrectomy and 12% perflouropropane (C3F8) gas tamponade and 20 patients Group 2 consisted of patients with epiretinal membrane or vitreous hemorrhage who underwent PPV without any tamponade
  Interventions: Other: pars plana vitrectomy

INTERVENTIONS:
Other: pars plana vitrectomy — 23 gauge pars plana vitrectomy was performed for retinal detachment, vitreous hemorrhage or epiretinal membrane

SUMMARY:
We aimed o compare the refractive changes associated with pars plana vitrectomy with or without intraocular gas tamponade in pseudophakic eyes. This retrospective study included pseudophakic patients with Nd:YAG laser posterior capsulotomy who underwent 23G PPV between February 2015 and March 2019. Group 1 consisted of patients with regmatogenous RD who underwent PPV and 12% perflouropropane (C3F8) gas tamponade whereas Group 2 consisted of patients who underwent PPV for epiretinal membrane or vitreous hemorrhage (VH). No tamponade was used in Group 2. Minimum follow-up was 12 months.

DETAILED DESCRIPTION:
This research was reviewed by an independent ethical review board and conforms with the principles and applicable guidelines for the protection of human subjects in biomedical research. This was a retrospective, comparative case series including pseudophakic patients who underwent PPV. Group 1 consisted of patients with pseudophakic RRD who underwent PPV and 12% perflouropropane (C3F8) gas tamponade whereas Group 2 consisted of patients with ERM or VH who underwent PPV without any tamponade between February 2015 and March 2019 at Bursa Retina Eye Hospital. Informed consent was obtained from all the participants. The study was in line with the ethical standarts of the Helsinki Declaration

Patient eligibility Patients who underwent uncomplicated cataract surgery with phacoemulsification and in-the-bag IOL implantation and subsequent neodymium:yttrium-aluminum-garnet (Nd:YAG) laser due to capsular opacification were included. Preoperative refractive data obtained after Nd:YAG laser and six months prior to vitrectomy surgery. Postoperative refractive data was obtained at 12 months after vitrectomy. Eyes with a preoperative spherical refractive error > ±6 D or cylindrical refractive error > ±3 D were excluded. Also eyes with corneal disorders were excluded.

Ocular parameters

All patients underwent complete ophtalmic examination including best corrected visual acuity (BCVA) in the logMAR scale, slit-lamp examination, intraocular pressure (IOP) assessment, fundus examination and autokeratorefractometry (auto kerato-refractometer KR-8800 from Topcon, Tokyo, Japan) at preoperative and postoperative month-12. Induced astigmatism values were calculated through vector analysis.

Surgical procedures

All surgeries were performed by the same surgeon (S.Y.). Retrobulbar block anesthesia (a mixture of 2 ml of lidocaine hydrochloride 2% and 2 ml of bupivacaine hydrochloride 0.5%) was used. Three port 23-gauge (G) transconjunctival PPV was performed using the vitrectomy system DORC (Dutch Ophthalmic Research Center, Zuidland, Netherlands) and Zeiss microscope with EIBOS 2 (Haag Streit, Mason, OH, USA) attachment for non-contact fundus viewing.

In group 1, all patients underwent a near-complete vitrectomy including base shaving, laser endo-photocoagulation and C3F8 gas tamponade. In group 2, patients with ERM received a limited vitrectomy including; core vitrectomy, induction of a posterior vitreous detachment if not present and peeling of the ERM and inner limiting membrane (ILM). Peripheral retina was examined with indentation to identify any retinal breaks. Neither laser endo-photocoagulation, nor gas tamponade and vitreous base shaving was performed. For patients with VH patients, a near-complete vitrectomy, including base shaving, laser endo-photocoagulation was performed except for gas tamponade. In both groups, the sclera is sutured with 8-0 polyglactin suture (Vicryl) in case of wound leakage.

ELIGIBILITY:
Inclusion Criteria

* Patients aged ≥ 18 years
* Pseudophakic patients who underwent pars plana vitrectomy

Exclusion Criteria

* Patients aged 18 years >
* Patients with a spherical refractive error > ±6 D
* Patients with a cylindrical refractive error > ±3 D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pseudophakic patients treated with neodymium:yttrium-aluminum-garnet Nd: YAG laser and subsequently underwent 23 gauge pars plana vitrectomy for vitreous hemorrhage, epiretinal membrane, or rhegmatogenous retinal detachment.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-27 (Actual)

PRIMARY OUTCOMES:
The rate of spherical and cylindrical refractive changes | 12 months
  Changes in spherical and cylindrical refractive error 12 months after pars plana vitrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Sami Yılmaz, MD, Principal Investigator — Bursa Retina Eye Hospital; Remzi Avcı, Professor, Study Director — Bursa Retina Eye Hospital; Aysegul Mavi Yıldız, MD, Principal Investigator — Bursa Retina Eye Hospital
Locations (1):
- Retina Eye Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hamoudi H, Kofod M, La Cour M. Refractive change after vitrectomy for epiretinal membrane in pseudophakic eyes. Acta Ophthalmol. 2013 Aug;91(5):434-6. doi: 10.1111/j.1755-3768.2012.02574.x. Epub 2012 Sep 23. PMID 22998208
- [Result] Byrne S, Ng J, Hildreth A, Danjoux JP, Steel DH. Refractive change following pseudophakic vitrectomy. BMC Ophthalmol. 2008 Oct 13;8:19. doi: 10.1186/1471-2415-8-19. PMID 18851731